CLINICAL TRIAL: NCT07157306
Title: Gecacitinib Combined With Donafenib and PD-1 Inhibitor as Second-Line Therapy for Unresectable Hepatocellular Carcinoma Failed in Immunotherapy, A Phase II Prospective Clinical Study
Brief Title: Gecacitinib Combined With Donafenib and PD-1 Inhibitor as Immune Rechallenge Therapy for Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Professor, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250854
Record Dates: First submitted 2025-08-14; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Immune re-challenge for HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): The participants in this arm will be treated with combination therapy of Gecacitinib（100mg,Bid,po）, Donafenib (200mg,Bid,po), and PD-1(Q3W,iv).
  Interventions: Drug: Gecacitinib Combined With Donafenib and PD-1 Inhibitor

INTERVENTIONS:
Drug: Gecacitinib Combined With Donafenib and PD-1 Inhibitor — Subjects were enrolled and started receiving treatment with Gecacitinib (100mg, Bid, po) for 7 consecutive days; thereafter, they were treated with PD-1 antibody (Q3W, iv) and Donafenib (200mg, Bid, po), counting the day of infusion of PD-1 monoclonal antibodies as C1D1, with each cycle lasting 3 weeks. Subsequent treatments involved administering Gecacitinib for 1 week before each infusion of PD-1.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Gecacitinib Combined With Donafenib and PD-1 Inhibitor as Immune Rechallenge Therapy for Unresectable Hepatocellular Carcinoma

DETAILED DESCRIPTION:
Jak inhibitors have already demonstrated the ability to reverse T-cell exhaustion in the treatment of Hodgkin lymphoma. Gecacitinib is a Jak inhibitor that has been approved for the treatment of bone marrow fibrosis. This study was designed to evaluate the safety and efficacy of Gecacitinib Combined With Donafenib and PD-1 Inhibitor as Immune Rechallenge Therapy for Unresectable Hepatocellular Carcinoma . Total 35 subjects will be recruited in this study, ORR will be will be used as primary outcome measures, OS, PFS, DCR and safety will be the secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: >18 years old and≤75 years old, both men and women.
2. All subjects must have Hepatocellular Carcinoma confirmed by pathological or clinical diagnosis.
3. Patients with viable and measurable target lesion per RECIST 1.1.
4. Patients with unresectable hepatocellular carcinoma (uHCC) who experienced disease progression after first-line therapy containing immune checkpoint inhibitors.
5. Patients who are expected to live more than 3 months.

9.ECOG PS 0-1. 10.Child-Pugh ≤7.

Exclusion Criteria:

1. Fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma confirmed by histology or cytology.
2. History of malignant tumor, excluding the following cases:

   1. Malignant tumor that was curatively treated more than 5 years prior to study entry and has not recurred since then;
   2. Successful radical resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, preinvasive cervix carcinoma, and other preinvasive cancers.
3. Diffuse tumor lesion.
4. Preexisting or history of hepatic encephalopathy, hepatorenal syndrome or liver transplantation.
5. Clinically uncontrolled ascites or pleural effusion.
6. Received treatment with a JAK inhibitor previously .
7. Clinically severe gastrointestinal bleeding within 6 months of the start of treatment or any life-threatening bleeding events within 3 months of the start of treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Evaluation of tumor burden based on mRECIST criteria

SECONDARY OUTCOMES:
OS | From date of enrollment until the date of death from any cause, assessed up to 3 years
PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Evaluation of tumor burden based on mRECIST criteria
DCR | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Evaluation of tumor burden based on mRECIST criteria
Incidence of treatment-related adverse events (TRAE) | From date of enrollment until the date of 30 days after the last treatment according to the protocol, assessed up to 3 years
  Number of patients with AE, treatment-related AE (TRAE), serious adverse event (SAE) assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathew D, Marmarelis ME, Foley C, Bauml JM, Ye D, Ghinnagow R, Ngiow SF, Klapholz M, Jun S, Zhang Z, Zorc R, Davis CW, Diehn M, Giles JR, Huang AC, Hwang WT, Zhang NR, Schoenfeld AJ, Carpenter EL, Langer CJ, Wherry EJ, Minn AJ. Combined JAK inhibition and PD-1 immunotherapy for non-small cell lung cancer patients. Science. 2024 Jun 21;384(6702):eadf1329. doi: 10.1126/science.adf1329. Epub 2024 Jun 21. PMID 38900877
- [Background] Zak J, Pratumchai I, Marro BS, Marquardt KL, Zavareh RB, Lairson LL, Oldstone MBA, Varner JA, Hegerova L, Cao Q, Farooq U, Kenkre VP, Bachanova V, Teijaro JR. JAK inhibition enhances checkpoint blockade immunotherapy in patients with Hodgkin lymphoma. Science. 2024 Jun 21;384(6702):eade8520. doi: 10.1126/science.ade8520. Epub 2024 Jun 21. PMID 38900864